CLINICAL TRIAL: NCT06907550
Title: Mitochondrial DNA Deletions in Plasma as a Diagnostic Aid for Females Presenting With Symptoms of Endometriosis
Status: Not yet recruiting | Type: Observational
Sponsor: Pearsanta, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: R2025-1001
Record Dates: First submitted 2025-03-27; First posted 2025-04-02 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Females suspected of endometriosis scheduled for laparoscopic surgery: Females suspected of endometriosis scheduled for laparoscopic surgery
  Interventions: Diagnostic Test: The Mitomic Endometriosis Test (MET) blood test for early detection of endometriosis

INTERVENTIONS:
Diagnostic Test: The Mitomic Endometriosis Test (MET) blood test for early detection of endometriosis — Patients will complete a questionnaire about their endometriosis symptoms and a sample of blood will be taken prior to their laparoscopy and sent to the laboratory for testing.

SUMMARY:
This study will investigate the clinical performance and diagnostic accuracy of the Mitomic® Endometriosis Test (MET) compared to laparoscopic diagnosis in a prospective clinical study in females presenting with symptoms suggestive of endometriosis. This study will recruit patients with suspected endometriosis who have been referred for a diagnostic laparoscopy. Patients will complete a questionnaire about their endometriosis symptoms and a sample of blood will be taken prior to their laparoscopy and sent to the laboratory for the MET to be run.

This study aims to first enroll 104 subjects to support the clinical validation necessary for launch of the test as an LDT. Following this, we plan a study extension with an aim to enroll up to 900 more (for a total of 1000) subjects to enable more precise estimation of performance characteristics, characterization of test performance in subtypes of endometriosis, to better understand the relationship between test results and secondary endpoints such as symptoms and demographic variables, and to establish a bank of samples to support future test development.

ELIGIBILITY:
Inclusion Criteria:

1. Be female, between menarche and menopause who present with symptoms of endometriosis at time of blood collection and are scheduled to undergo their first laparoscopic procedure for the diagnosis of endometriosis
2. Provide a blood sample prior to surgical procedure or administration of drugs related to the surgical procedure (i.e. anaesthetics, antibiotics)
3. Be fit to undergo all procedures listed in protocol
4. Be able to provide written informed consent

Exclusion Criteria:

1. Has had a prior surgical diagnosis of endometriosis at time of blood collection
2. Is unable to communicate in written and spoken English
3. Has any other condition, which in the opinion of the investigator, would make the subject not a suitable candidate for the study. This reason must be recorded on the CRF

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Females between menarche and menopause presenting with symptoms suggestive of endometriosis and scheduled for a standard-of-care diagnostic laparoscopy
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of endometriosis | up to 5 years
  Presence or absence of endometriosis as determined by standard-of-care diagnostic laparoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Varvel, Ph.D., Principal Investigator — Pearsanta, Inc
Locations (1):
- Pearsanta, Inc., Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided